CLINICAL TRIAL: NCT05573633
Title: Diagnosis of Postoperative Atrial Fibrillation After Cardiac Surgery by a Smartwatch: an Open-label Randomized Controlled Trial
Brief Title: Diagnosis of Postoperative Atrial Fibrillation by a Smartwatch
Acronym: FAWATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI2021_843_0228
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: smartwatch; Atrial Fibrillation; perioperative atrial fibrillation; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smartwatches group (Experimental)
  Interventions: Procedure: scanwatch
- no smartwatche group (Active Comparator)
  Interventions: Procedure: ECG

INTERVENTIONS:
Procedure: ECG — the POAF will be diagnosed using a 12-lead ECG and according to the usual monitoring protocols for patients in the cardiac surgery department of Amiens University Hospital.
  Arms: no smartwatche group
Procedure: scanwatch — POAF will be diagnosed with a Withings SM (ScanWatch). FAPO diagnosed by the SW will have to be confirmed by a 12-lead ECG.
  Arms: smartwatches group

SUMMARY:
The incidence of postoperative atrial fibrillation (POAF) after on-pump cardiac surgery remains high, at around 30%. POAF increases the risk of cardiac decompensation, stroke, acute myocardial infarction, and death, resulting in increased morbidity and mortality, hospital length of stay, and cost of patient management. Episodes of POAF are usually paroxysmal and asymptomatic, increasing the risk of developing permanent AF at five years by 4 to 5 times. POAF occurs between 3 and 4 days after cardiac surgery, mainly when the patient is hospitalized in a surgical ward without heart rate monitoring as opposed to critical care, where the patient benefits from continuous rhythmic monitoring. The diagnosis of POAF is therefore made with the help of a 12-lead electrocardiogram (ECG) when the patient presents clinical symptoms and when the medical staff notes a significant variation in heart rate. However, many patients with episodes of asymptomatic POAF have a higher risk of stroke and mortality than those with symptomatic POAF.

Faced with this public health problem, the development of tools for diagnosing AF is in full swing, mainly the marketing of smartwatches (SWs) that allow for the performance of 1-lead ECG. SW is also equipped with algorithms to analyze heart rate variability and diagnose asymptomatic atrial fibrillation (AF) episodes. The European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS) recommend the use of smartwatches to detect AF, in particular, to reduce the economic impact of AF.

The aim of the study is to diagnose POAF within the first five days after patient discharge from the critical care unit for the cardiac surgery department.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years old)
* The patient was hospitalized at Amiens University Hospital for on-pump cardiac surgery.
* The patient has had a recent on-pump cardiac surgery (< 96h)
* Patient with the motor and cognitive abilities to perform a 1-lead ECG with the smartwatch
* The patient was transferred to the cardiac surgery department of Amiens University Hospital.
* The beneficiary of a social security plan
* Signature of the consent to participate in the study

Exclusion Criteria:

* History of AF
* Need for rhythmic monitoring by telemetry in cardiac intensive care for atrioventricular block and rapid supra and ventricular rhythm disorder (>140 bpm).
* An external pacemaker connected to epicardial electrodes depends on ventricular and atrial pacing.
* Patients already included in an interventional clinical research protocol may alter the incidence of POAF.
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2028-07-06 (Estimated)

PRIMARY OUTCOMES:
Variation of POAF incidence between both groups | 5 days
  The incidence of POAF will be compared between the two arms

SECONDARY OUTCOMES:
percentage of asymptomatic POAF in the SW arm | 5 days
Association between POAF and left atrial reservoir strain | At the enrollment in the study (day 0)
  Left atrial reservoir strain (LASr), measured by transthoracic echocardiography at discharge from the cardiothoracic intensive care unit to the conventional ward, expressed as a percentage (%), and analyzed for its association with POAF (comparison between patients with and without POAF).
Feasibility of rhythm monitoring using a smartwatch | 5 days
  The feasibility of rhythm monitoring using a smartwatch will be assessed by wear time of the smartwatch during the protocol period
Cardiovascular prognosis assessed by the occurrence of major adverse cardiovascular events (MACE) | 3 months and 6 months after inclusion
  Cardiovascular prognosis will be assessed using a composite endpoint of postoperative cardiovascular complications (MACE), defined according to the standards of the European Society of Anaesthesiology (ESA). MACE will be considered present if at least one of the following events occurs: stroke; Myocardial infarction; Digestive ischemia; Unplanned hospitalization for acute right and/or left heart failure decompensation; Resuscitated cardiac arrest and Cardiovascular death.
  Unit : Frequency of patients experiencing at least one MACE event (percentage, %).
Percentage of patients POAF after hospital discharge. | 3 months and 6 months
  Percentage of patients with POAF after hospital discharge in both groups (with and without smartwatch), assessed at 3 and 6 months after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No